CLINICAL TRIAL: NCT05466903
Title: Early Diet Opening on Postoperative Gastrointestinal Hemorrhage in Patients With Colonic Polyps
Brief Title: Prospective, Randomized, Parallel Clinical Controlled Study of Early Diet Opening on Postoperative Gastrointestinal Hemorrhage in Patients With Colonic Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Yan2020-204
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Colonic Polyp
Keywords: Colonic Polyp; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Colonic Polyps; Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): patients were given a liquid diet 6 hours after the operation
- Experimental arm (Experimental): patients were given a liquid diet 2 hours after the operation
  Interventions: Dietary Supplement: Early diet opening

INTERVENTIONS:
Dietary Supplement: Early diet opening — Effects of early dietary recovery after colon polypectomy and colonoscopic mucosal resection on postoperative hemorrhage in patients
  Arms: Experimental arm

SUMMARY:
Currently, hemorrhage remains the most common postoperative complication in patients with colon polyps, with an incidence of approximately 1.5%. The main reasons for postoperative hemorrhage are: the patient's own condition, the nature of the polyp and the operation. The number of patients treated for colon polyps has increased, postoperative care is confusing, medical resources are wasted, and the time span for postoperative diet recovery is large. However, studies on the effect of postoperative dietary recovery timing on postoperative polyp bleeding are rare.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, no gender restrictions,
* Patients with colonic polyps identified by colonoscopy and requiring endoscopic treatment,
* Polyp size 0.5cm-2cm,
* Patients agreed to enroll and signed a written informed consent,
* Adherence is good and agrees to be treated and evaluated as required by the study protocol.

Exclusion Criteria:

* Patients with contraindications to endoscopic treatment of colonic polyps, including platelets ≤50×109/L, prothrombin time prolonged by 4 seconds or more, and INR≥2.0,
* Patients with severe heart, brain, lung, blood system diseases, uremia, connective tissue disease,
* Patients requiring treatment with NSAIDs, aspirin, glucocorticoids, or clopidogrel within the first 7 days of the study,
* During the course of the study, due to other concomitant/complications, patients who need to use drugs that affect the efficacy of the trial, including various anticoagulants, antiplatelet drugs and hemostatic drugs,
* Alcoholics, drug addicts or those with uncontrollable neuropsychiatric diseases and others who are not suitable for participating in the trial,
* Pregnant, breastfeeding women, or women in childbearing age who wish to become pregnant,
* Patients with malignant tumor of digestive system,
* Other circumstances in which the investigator believes that the patient should not participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative bloody stool | up to 2 weeks
  Postoperative massive hemorrhage: if the amount of blood in stool exceeds 400ml within 1 hour to 14 days after operation, or the hemoglobin decreases >2g/dl
  Ordinary hemorrhage: the amount of blood in stool does not meet the above standards

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, the 2nd Affiliated Hospital of Medical College, Zhejiang University, Hangzhou, Zhejiang, China